CLINICAL TRIAL: NCT05757843
Title: Using Circulating Tumor DNA to Personalize Duration of Consolidation Durvalumab in Patients with Inoperable Stage III Non-small Cell Lung Cancer: the Indiana Trial
Brief Title: Using Circulating Tumor DNA to Personalize Duration of Consolidation Durvalumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to identify patients who meet eligibility requirements of tissue needed for analysis.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nasser Hanna, Tom and Julie Wood Family Foundation Professor of Lung Cancer Clinical Research, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0749
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NSCLC, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Consolidation to Durvalumab (Experimental): All subjects will receive consolidation Durvalumab approximately every 4 weeks. The first mandatory ctDNA test will be done at screening for the bespoke ctDNA profiling. The next mandatory ctDNA test will be completed prior to the 5th cycle of consolidation Durvalumab. If it's negative and the subsequent test 4 weeks later prior to cycle 6 is negative, then Durvalumab will be stopped otherwise subject will continue consolidation durvalumab until 2 negative ctDNA analyses performed approximately 4 weeks apart or up to 1 year of consolidation per standard medical practice is complete.
  Interventions: Diagnostic Test: Signatera ctDNA test; Drug: Durvalumab

INTERVENTIONS:
Diagnostic Test: Signatera ctDNA test — The first mandatory ctDNA test will be done at screening for the bespoke ctDNA profiling. The next mandatory ctDNA test will be completed prior to the 5th cycle of consolidation Durvalumab. ctDNA testing will be repeated approximately every 4 weeks until two consecutive negative analyses occur. ctDNA testing will be otherwise discontinued after progressive disease or after up to 1 year of consolidation treatment per standard medical practice is considered complete, whichever occurs first.
Drug: Durvalumab — All subjects will receive consolidation Durvalumab approximately every 4 weeks. Durvalumab will be stopped after two consecutive negative ctDNA analyses occur.

SUMMARY:
This research aims to incorporate ctDNA analysis into clinical practice to individualize therapy in patients with stage III NSCLC by moving to a treatment-by-marker based approach (as opposed to treatment based on clinical or radiographic evidence of disease).

DETAILED DESCRIPTION:
There is a critical need to identify MRD to determine which patients benefit from checkpoint inhibitor therapy and to optimize and personalize the duration of consolidation Durvalumab. The long-term goal is to incorporate ctDNA analysis into clinical practice to individualize therapy in patients with stage III NSCLC by moving to a treatment-by-marker based approach (as opposed to treatment based on clinical or radiographic evidence of disease). This approach may spare a subset of patients from treatment with unnecessarily excessive cycles of consolidation immunotherapy if they are already cured with CRT alone and individualize the duration of consolidation immunotherapy in patients not cured with CRT. The study team also seek to identify early in the treatment course, patients who are destined not to be cured with consolidation immunotherapy so that alternative strategies can be tested when tumor burden is low.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Ability to provide written informed consent and HIPAA authorization

Patients with inoperable or unresectable stage III NSCLC who are planning to receive concurrent CRT followed by consolidation Durvalumab OR Patients with inoperable or unresectable stage III NSCLC who have previously received concurrent CRT and are planning or currently receiving C1-4 consolidation durvalumab

Must have viable tissue for ctDNA profiling, (fresh or archived tissue)

Exclusion Criteria:

Patient unwilling to provide tissue and blood samples for ctDNA testing.

Patient has contraindications to treatment with concurrent CRT and/or consolidation Durvalumab.

Patients with any other active cancer; excluding squamous cell or basal cell cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine if de-escalating number of Durvalumab cycles based on personalized ctDNA clearance has non-inferior 2-year PFS rate | Baseline to 24 months
  Determine if de-escalating the number of Durvalumab cycles based on personalized ctDNA clearance guidance to at least 6 cycles after CRT in stage III non-resectable NSCLC has non-inferior 2-year PFS rate compared with historical control of empirically treating stage III non-resectable NSCLC for 1 year of Durvalumab after CRT.

SECONDARY OUTCOMES:
Estimate the 24-month overall survival (OS) of patient treated with consolidation Durvalumab based on personalized ctDNA clearance | Baseline to 24 months
  Estimate the 24-month overall survival (OS) of patient treated with consolidation Durvalumab based on personalized ctDNA clearance guidance for at least 6 cycles after CRT in stage III non-resectable NSCLC.
Estimate the 24-month PFS in patients with persistently detectable ctDNA without radiographic progression | Baseline to 24 months
  Estimate the 24-month PFS in patients with persistently detectable ctDNA without radiographic progression of disease after receiving ≥ 6 months of consolidation Durvalumab.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University